CLINICAL TRIAL: NCT02262507
Title: Concussion Device Audiological Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-5717
Record Dates: First submitted 2014-10-03; First posted 2014-10-13 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Concussion; Traumatic Brain Injury
Keywords: Brain; Hearing; MTBI
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device wearing (Experimental): All subjects who meet the study criteria and volunteer to participate will be included in the study. Subjects will undergo repeat oto-acoustic measures both wearing the device and not wearing the device. The intervention will be the auto-acoustic measurement - taken while wearing the collar and then again when not wearing the collar.
  Interventions: Device: Device Wearing

INTERVENTIONS:
Device: Device Wearing — Q30 collar - collar designed to be worn around the neck to apply slight pressure to jugular veins. Each subject will undergo repeat oto-acoustic measures both wearing the device and not wearing the device

SUMMARY:
Significant morbidity, mortality, and related costs are caused by traumatic brain injury (TBI). A simple, effective, and lightweight device worn by athletes or war fighters in the field, designed to mitigate TBI resulting from blast trauma or concussive events, would save lives, and the huge costs currently being experienced for life-treatment of surviving victims. An externally-worn medical device that applies mild jugular compression according to the principle of the Queckenstedt Maneuver (the Device) is being developed by Q30 Labs, LLC (Q30). Initial research suggests that the Device has the potential to reduce the likelihood of TBI. The rationale for testing wideband absorbance and Oto-acoustics emissions (OAE) is that the investigators need a physiologic, non-invasive method to evaluate the brain responses to mild jugular compression across multiple age groups. To determine this with MR imaging is currently cost prohibitive. The investigators pilot data from the parent IRB indicates a consistent response measured via wideband absorbance in young adults. Therefore, a preliminary step to evaluate the safety and efficacy of the neck collar device is to employ this technology across a wide range of ages.

DETAILED DESCRIPTION:
For the testing sessions, subjects may either come to our testing site or the investigators may bring the testing to their location (e.g. schools, work). The subjects will be fitted with a device around your neck, like a neck tie. The Device incorporates two bulges localized over the site of the internal jugular veins bilaterally. Experiments performed with jugular Doppler ultrasound demonstrate that while wearing the Device, flows within the jugular veins are reduced, while flow within the carotid arteries and all portions of the cerebrum are preserved (JA Fisher, unpublished data). Thus, application of the Device to the subject will not cause any untoward health risks (IRB# 2013-2240 safety testing performed on this Device). The pressure exerted by the Device on the region of the neck superficial to the internal jugular vein is akin to the pressure felt when a person yawns or wears a snugly fitting necktie. The methods are utilized in prior approved IRB (2013-2240)..

Station I: Consent to Participate Each participant will review the Institutional Review Board approved consent to participate form prior to data collection. They will be given an adequate amount of time to ask questions to the study coordinator, or the person obtaining consent, and then make their decision to participate or not participate. If they wish to participate, they will be asked to sign the informed consent form. For middle school and high school subjects recruited via the investigators relationship with the schools, this station will be designated to review consent and assent forms to ensure that proper signatures have been obtained.

Station II: Device Fitting and Ultrasound The subjects will be outfitted with the device by a staff member appropriately trained in fitting the device in the proper location.

Station III: Wideband Absorbance and Oto-Acoustic Emissions This station will help determine the effectiveness of the device by measuring the auditory response of a clicking noise that will be non-invasively imparted into the subject's outer ear. For both tests, a soft silicone tip is placed into the outer ear, and sounds are delivered via a miniature speaker. For the wideband absorbance test, absorbed acoustic responses will be monitored to provide information on the operation of the collar device. These are measured as changes in the acoustic absorbance of the ear. For the oto-acoustic emission test, tones or clicks will be presented to the ear with the same soft ear probe and recording microphones pick up the oto-acoustic emission coming back from the outer hair cells of the inner ear. The computer averages and processes the responses in reference to a noise floor across a specified frequency range, displaying the results on the computer screen for the tester. The oto-acoustic emissions test also provides a brief hearing screening to determine if hearing is normal.

Evidence indicates that wideband absorbance and oto-acoustic emissions will be altered with increased intracranial pressure, thus this simple, non-invasive exam will provide feedback on the effectiveness of the device.

During the wideband absorbance and oto-acoustic emissions testing the study participants will also be fitted with a compressive circumferential neck collar which can provide variable and specific levels of pressure. The pressure is achieved by inflatable pods that sit adjacent to the trachea affixed to a non-stretch adjustable collar. Manual inflation is regulated and monitored by an experience operator/ technician through a bulb style pump and an electronic gauge. Testing will occur without pressure and then with pressures applied up to 40mmHg.

Station IV: Hearing Assessment Otoscopy will be performed by an audiologist to note any ear blockages, such as wax or drainage for exclusion purposes. The oto-acoustic emissions test will be interpreted to determine if normal responses were obtained in each ear. If abnormal, a hearing screening using pure tone audiometry screening will be provided free of charge. In the event that the hearing screening is determined to be abnormal, the subject will receive the results which may be shared with their primary care provider to determine any need for referral for follow-up. If a subject is seen for follow-up at CCHMC following an abnormal hearing assessment, this visit and any follow up visits will not be paid for by this project and will be subject to insurance billing.

ELIGIBILITY:
Inclusion Criteria:

* • Normal healthy volunteer

  * Able to provide written consent

Exclusion Criteria:

* • Unable to provide written consent

  * History of neurological deficits, previous cerebral infarction, or head trauma
  * Hydrocephalus
  * Known carotid hypersensitivity
  * Known increased intracranial pressure
  * Central vein thrombosis
  * Active concussion symptoms
  * Ventricular shunt or neurologic condition
  * Internal or external hardware that has been surgically placed in the neck
  * Any altered level of consciousness
  * Inability to sit still for 10 minutes

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

RESULTS

PARTICIPANT FLOW:
Groups:
- Device Wearing: All subjects who meet the study criteria and volunteer to participate will be included in the study.
  Q Collar: Q30 collar - collar designed to be worn around the neck to apply slight pressure to jugular veins. subjects will undergo repeat oto-acoustic measures both wearing the device and not wearing the device.
Period: Overall Study
Arm/Group | Device Wearing
Started | 410
Completed | 410
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Device Wearing: All subjects who meet the study criteria and volunteer to participate will be included in the study.
  Q Collar: Q30 collar - collar designed to be worn around the neck to apply slight pressure to jugular veins
Arm/Group | Device Wearing
Number analyzed (Participants) | 410
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 335
  Between 18 and 65 years | 74
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 18.5 [12 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251
  Male | 159
Region of Enrollment [Number; unit: participants]
  United States | 410

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Undergoing Acoustic Reflectance
Description: Number of participants undergoing acoustic reflectance with and without the compression collar
Time Frame: within single day
Population: Subjects
Measure: Number; unit: participants
Groups:
- Non Device Wearing: same subjects tested while not wearing the device
Arm/Group | Device Wearing | Non Device Wearing
Number analyzed (Participants) | 410 | 410
participants | 410 | 410
Statistical Analysis 1: Comparison: Device Wearing; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- Device Wearing: All subjects who meet the study criteria and volunteer to participate will be included in the study.
  Q Collar: Q30 collar - collar designed to be worn around the neck to apply slight pressure to jugular veins Subjects will undergo repeat oto-acoustic measures both wearing the device and not wearing the device.
Arm/Group | Device Wearing
Serious Adverse Events (participants affected / at risk) | 0/410
Other Adverse Events (participants affected / at risk) | 0/410

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-10-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT02262507/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT02262507/ICF_001.pdf